CLINICAL TRIAL: NCT00920699
Title: A Multi-Center, Double-Blind, Randomized, Parallel Group Tolerability Study of Coenzyme Q10 (UbiquinonE)in PRE-manifest Huntington's Disease
Brief Title: Study in PRE-manifest Huntington's Disease of Coenzyme Q10 (UbiquinonE) Leading to Preventive Trials (PREQUEL)
Acronym: PREQUEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PREQUEL-01.00; NIH grant: 1 R01 NS060118-01A1
Record Dates: First submitted 2009-06-09; First posted 2009-06-15 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 600 mg per day of CoQ10 (Experimental): All participants will start on a dosage of 600 mg/day of CoQ10 in divided doses, increasing weekly by 600 mg/day to a maximum dosage of 2400 mg/day at week 4. Dosage should be stable from week 4 until week 20.
  Interventions: Drug: CoQ10
- 1200 mg per day of CoQ10 (Experimental): All participants will start on a dosage of 600 mg/day in divided doses, increasing weekly by 600 mg/day to a maximum dosage of 2400 mg/day at week 4. Dosage should be stable from week 4 until week 20.
  Interventions: Drug: CoQ10
- 2400 mg per day of CoQ10 (Experimental): All participants will start on a dosage of 600 mg/day in divided doses, increasing weekly by 600 mg/day to a maximum dosage of 2400 mg/day at week 4. Dosage should be stable from week 4 until week 20.
  Interventions: Drug: CoQ10

INTERVENTIONS:
Drug: CoQ10 — Capsules containing 300 mg of CoQ10 or matching placebo taken orally twice a day. All participant will start on a dosage of 600 mg/day in divided doses, increasing weekly by 600 mg/day to a maximum dosage of 2400 mg/day at week 4. Dosage should be stable from week 4 until week 20.
  Other Names: -Ubiquinone; -coenzyme Q10

SUMMARY:
To establish the tolerability of treatment with 600, 1200 or 2400 mg per day of coenzyme Q10 in pre-manifest participants carrying the CAGn expansion for Huntington's Disease (HD).

DETAILED DESCRIPTION:
secondary objectives:

1. To assess the change from baseline to 20 weeks on biomarkers of oxidative stress (8OHdG and 8OHrG) and DNA repair mechanisms (OGG1) in pre-manifest participants treated with 600, 1200 or 2400 mg per day of CoQ10.
2. To assess the dose-response relationship between CoQ10 at dosages of 600, 1200 or 2400 mg per day and 8OHdG/8OHrG and OGG1.
3. To assess the serum levels of CoQ10 at 600, 1200 or 2400 mg in pre-manifest participants and their relationship to 8OHdG/8OHrG and OGG1.
4. To assess the feasibility of implementing a preventive therapeutic trial in a pre-manifest population.
5. To assess the utility and stability of clinical measures of HD, social relations, behavior and employment in a pre-manifest sample enrolled in a treatment trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be positive for the CAGn expansion in the Huntingtin gene (>36 repeats) and be pre-manifest by virtue of scoring 3 or less on diagnostic confidence level (Question 17 of the UHDRS)
* Participants will have received genetic testing prior to enrollment through a standard pre-manifest testing protocol.
* 18 years of age or older.
* Concomitant medications are permitted with the exception of CoQ10, creatine > 5g/day and warfarin.

Exclusion Criteria:

* History of intolerability to CoQ10.
* CoQ10 use within 60 days prior to randomization.
* Unstable medical or psychiatric illness;
* Substance abuse within one year of the baseline visit.
* Pregnancy, breastfeeding or lack of reliable contraception in women of childbearing age.
* Subjects with known allergy to FD&C #6 yellow food coloring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Ross, MD, PhD, Principal Investigator — Johns Hopkins University; Kevin M Biglan, MD, MPH, Principal Investigator — University of Rochester
Locations (13):
- United States (13):
  - University of California Davis, Sacramento, California
  - Colorado Neurological Institute, Englewood, Colorado
  - University of Miami School of Medicine, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Hereditary Neurological Disease Centre (HNDC), Wichita, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - University of Rochester, Rochester, New York
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- See also: Huntington Study Group — http://www.huntington-study-group.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 600 mg Per Day of CoQ10 | 1200 mg Per Day of CoQ10 | 2400 mg Per Day of CoQ10
Started | 29 | 30 | 32
Completed | 27 | 29 | 28
Not Completed | 2 | 1 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — no longer met eligibility | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: one subject no longer met eligibility criteria in the 1200 mg arm
Groups:
- Total: Total of all reporting groups
Arm/Group | 600 mg Per Day of CoQ10 | 1200 mg Per Day of CoQ10 | 2400 mg Per Day of CoQ10 | Total
Number analyzed (Participants) | 29 | 29 | 32 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (9.8) | 39.3 (11.5) | 39.8 (11.6) | 39.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 16 | 47
  Male | 14 | 13 | 16 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 29 | 32 | 90

OUTCOME MEASURES:

1. Primary Outcome: Tolerability as Assessed by Ability to Complete the Study on the Originally Randomized Treatment Assignment.
Description: No dosage modifications, reported as a %
Time Frame: 20 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 600 mg Per Day of CoQ10 | 1200 mg Per Day of CoQ10 | 2400 mg Per Day of CoQ10
Number analyzed (Participants) | 29 | 29 | 32
percentage of participants | 90.0 | 93.1 | 81.3

2. Secondary Outcome: 8OHdG Levels
Description: ng/ml. Negative value signifies an decrease in 8OHdG levels
Time Frame: change from baseline to 20 weeks
Population: Lab data not available for all participants to compare baseline and 20 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 600 mg Per Day of CoQ10 | 1200 mg Per Day of CoQ10 | 2400 mg Per Day of CoQ10
Number analyzed (Participants) | 19 | 21 | 27
ng/ml | 0.15 (3.26) | -1.56 (3.23) | 0.55 (7.1)

3. Secondary Outcome: CoQ10 Levels
Description: ng/ml
Time Frame: change from baseline to 20 weeks
Population: data was not available for all participants to compare baseline to 20 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 600 mg Per Day of CoQ10 | 1200 mg Per Day of CoQ10 | 2400 mg Per Day of CoQ10
Number analyzed (Participants) | 24 | 25 | 28
ng/ml | 1.82 (1.78) | 1.92 (1.66) | 2.33 (1.38)

ADVERSE EVENTS:
Time Frame: up to 20 weeks
Arm/Group | 600 mg Per Day of CoQ10 | 1200 mg Per Day of CoQ10 | 2400 mg Per Day of CoQ10
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 9/29 | 20/29 | 16/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600 mg Per Day of CoQ10 (N=29) | 1200 mg Per Day of CoQ10 (N=29) | 2400 mg Per Day of CoQ10 (N=32)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 7 (7) | 4 (4)
Abdominal discomfort/pain; dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
increase creatinine phosphokinase (blood) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes